| Role of Mirtazapin | e in / | Ameliorating | Sleep | <b>Disordered</b> | <b>Breathing</b> |
|---|---|---|---|---|---|

NCT04799782 Abdulghani Sankari, MD, PhD 4/14/2021 Statistical Analysis: Demographic characteristics (age, gender, BMI and level of SCI injury) are summarized as mean and standard deviation (SD) or frequency and percentage scores, as applicable. A paired-samples t-test is used to examine the change in CO2 reserve (primary outcome), CG, plant gain (PG), as well as SDB and ventilatory parameters (secondary outcomes) between the two treatment groups (Mirtazapine vs. placebo). The SDB parameter include apnea-hypopnea index, sleep staging and timing, oxygen desaturation index and arousal index. The ventilatory parameters include tidal volume, frequency and minute ventilation. All analyses are considered as statistically significant at p≤ 0.05.